CLINICAL TRIAL: NCT05765773
Title: An Open Comprative Study of the Prophylactic Efficacy and a Non-comparative Study of the Immunogenicity and Safety of the Inactivated Whole-virion Concentrated Purified Coronavirus Vaccine (CoviVac) for Adults Aged 60 Years and Older
Brief Title: An Open Comparative Study of the Effectiveness and Incomparable Study of the Immunogenicity and Safety of the Vaccine (CoviVac) for Adults Aged 60 Years and Older
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chumakov Federal Scientific Center for Research and Development of Immune-and-Biological Products (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: № VKI-P-II-07/21
Record Dates: First submitted 2023-02-13; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-02

CONDITIONS: Corona Virus Infection; Vaccine; COVID-19
Keywords: COVID-19; SARS-Cov-2
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The study group consisted of 200 volunteers (Experimental): The study group is planned to screen a maximum of 250 volunteers inclusive, of which it is planned to include 200 men and women aged 60 years and older who meet the criteria for inclusion in the study and do not have non-inclusion criteria.
  Interventions: Biological: CoviVac vaccine (inactivated whole-virion concentrated purified) manufactured by FSBSI "Chumakov FSC R&D IBP RAS"
- Control group (No Intervention): Retrospective immunogenicity data obtained in the framework of clinical study № VKI-I/II-08/20 on healthy volunteers aged 18-60 years.

INTERVENTIONS:
Biological: CoviVac vaccine (inactivated whole-virion concentrated purified) manufactured by FSBSI "Chumakov FSC R&D IBP RAS" — 200 volunteers who will be vaccinated with the CoviVac vaccine three times with an interval of 21 days intramuscularly at a dose of 0.5 ml.
  Arms: The study group consisted of 200 volunteers

SUMMARY:
An Open Comprative Study of the Prophylactic Efficacy and a Non-comparative Study of the Immunogenicity and Safety of the Inactivated Whole-virion Concentrated Purified Coronavirus Vaccine (CoviVac) Produced by FSBSI "Chumakov Federal Scientific Center for Research and Development of Immune-and-Biological Products" for Adults Aged 60 Years and Older

DETAILED DESCRIPTION:
An open comparative multicenter prospective study with retrospective data.

ELIGIBILITY:
Inclusion Criteria:

Volunteers must meet the following inclusion criteria:

Type of participants

• Healthy volunteers or volunteers with a history of stable diseases that do not meet any of the criteria for non-inclusion in the study.

Other inclusion criteria

* Written informed consent of volunteers to participate in a clinical trial
* Volunteers who are able to fulfill the Protocol requirements (i.e., fill out a self-observation Diary, come to control visits).

Exclusion Criteria:

SARS-CoV-2 infection • A case of established COVID-19 disease confirmed by PCR and/or ELISA in the last 6 months.

Diseases or medical conditions

* Serious post-vaccination reaction (temperature above 40 C, hyperemia or edema more than 8 cm in diameter) or complication (collapse or shock-like condition that developed within 48 hours after vaccination; convulsions, accompanied or not accompanied by a feverish state) to any previous vaccination.
* Burdened allergic history (anaphylactic shock, Quincke's edema, polymorphic exudative eczema, serum sickness in the anamnesis, hypersensitivity or allergic reactions to the introduction of any vaccines in the anamnesis, known allergic reactions to vaccine components, etc.).
* Guillain-Barre syndrome (acute polyradiculitis) in the anamnesis.
* The axillary temperature at the time of vaccination is more than 37.0 ° C.
* Acute infectious diseases (recovery earlier than 4 weeks before vaccination) according to anamnesis.
* Donation of blood or plasma (in the amount of 450 ml or more) less than 2 months before inclusion in the study.
* Severe and/or uncontrolled diseases of the cardiovascular, bronchopulmonary, neuroendocrine systems, gastrointestinal tract, liver, kidneys, hematopoietic, immune systems.
* Is registered at the dispensary for tuberculosis, leukemia, oncological diseases, autoimmune diseases.
* Any confirmed or suspected immunosuppressive or immunodeficiency condition in the anamnesis.
* Splenectomy in the anamnesis.
* Neutropenia (decrease in the absolute number of neutrophils less than 1000/mm3), agranulocytosis, significant blood loss, severe anemia (hemoglobin less than 80 g/l) according to anamnesis.
* Anorexia according to anamnesis.

Prior or concomitant therapy

* Vaccination with any vaccine carried out within 30 days before vaccination / the first dose of the studied vaccine or planned administration within 30 days after vaccination / the last dose of the studied vaccine.
* Prior vaccination with an experimental or registered vaccine that may affect the interpretation of the study data (any coronavirus or SARS vaccines).
* Long-term use (more than 14 days) of immunosuppressants or other immunomodulatory drugs (immunoregulatory peptides, cytokines, interferons, immune system effector proteins (immunoglobulins), interferon inducers (cycloferon) during the six months preceding the study, according to anamnesis.
* Treatment with systemic glucocorticosteroids (≥ 20 mg of prednisone, or an analog, for more than 15 days during the last month).
* Volunteers who received immunoglobulin preparations or blood transfusion during the last 3 months prior to the start of the study according to anamnesis.

Other non-inclusion criteria

• Participation in any other clinical trial within the last 3 months.

Exclusion criteria:

* Withdrawal of Informed consent by a volunteer;
* The volunteer was included in violation of the inclusion/non-inclusion criteria of the Protocol;
* Any condition of a volunteer that requires, in the reasoned opinion of a medical researcher, the withdrawal of a volunteer from the study;
* Taking unauthorized medications (see section 6.2);
* The volunteer refuses to cooperate or is undisciplined (for example, failure to attend a scheduled visit without warning the researcher and/or loss of communication with the volunteer), or dropped out of observation;
* For administrative reasons (termination of the study by the Sponsor or regulatory authorities), as well as in case of gross violations of the Protocol that may affect the results of the study.

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of development, type and association with vaccination of adverse events during the study. | 6 month
  Frequency of development, type and association with vaccination of adverse events during the study.
Titer of specific antibodies | 21 days
  The proportion of volunteers from the total number of vaccinated with the level of seroconversion (titer of specific antibodies = 4 times the baseline level) on 21 days after the course of vaccination in the reaction of viral neutralization and / or ELISA.
GMT on day 21 after the course of vaccination | 21 days
  The proportion of volunteers with an increase in the level of immune response in the form of geometric mean titers of specific antibodies (GMT) on day 21 after the course of vaccination in the reaction of viral neutralization and / or ELISA.
The frequency of occurrence of clinically significant deviations from the norm of the main indicators of vital functions and laboratory parameters. | 6 month
  The frequency of occurrence of clinically significant deviations from the norm of the main indicators of vital functions and laboratory parameters.

SECONDARY OUTCOMES:
ARVI, COVID-19 | 6 month
  Frequency, severity and duration of incidence of Acute respiratory diseases (ARVI, COVID-19) within six months after triple vaccination.

CONTACTS AND LOCATIONS:
Locations (7):
- Russia (7):
  - State Budgetary Healthcare Institution of the Moscow region "Elektrostal Central City Hospital", Elektrostal, Moscow Oblast
  - Federal State Budgetary Scientific Institution "I.I. Mechnikov Scientific Research Institute of Vaccines and Serums", Moscow
  - FSBSI Chumakov FSC R&D IBP RAS, Moscow
  - Private healthcare institution "Clinical Hospital "Russian Railways-Medicine" named after N.A. Semashko", Moscow
  - Limited Liability Company "Scientific Research Center Ecosecurity", Moscow
  - Federal State Budgetary Healthcare Institution "Medical and Sanitary Unit No. 163 of the Federal Medical and Biological Agency", Novosibirsk
  - Federal State Budgetary Educational Institution of Higher Education "Perm State Medical University named after Academician E.A. Wagner" of the Ministry of Health of the Russian Federation, Perm